CLINICAL TRIAL: NCT04064242
Title: A Subject and Investigator Blinded, Randomized, Placebo-controlled, Repeat-dose, Multicenter Study to Investigate Efficacy, Safety, and Tolerability of CMK389 in Patients With Chronic Pulmonary Sarcoidosis
Brief Title: Study of Efficacy, Safety and Tolerability of CMK389 in Patients With Chronic Pulmonary Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCMK389X2201
Record Dates: First submitted 2019-08-20; First posted 2019-08-21 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Sarcoidosis
Keywords: chronic pulmonary sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two treatment arms, either CMK389 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CMK389 (Experimental): CMK389 10 mg/kg i.v. every 4 weeks for a total of 4 doses
  Interventions: Drug: CMK389
- Placebo (Placebo Comparator): Placebo i.v. every 4 weeks for a total of 4 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CMK389 — single i.v. dose every 4 weeks
  Arms: CMK389
Drug: Placebo — single i.v. dose every 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this proof of concept study was to determine whether CMK389 displays the safety and efficacy profile to support further development in chronic pulmonary sarcoidosis.

DETAILED DESCRIPTION:
This was a subject and investigator blinded, randomized, placebo-controlled, parallel-group, repeat-dose, multicenter, non-confirmatory study of CMK389 in chronic pulmonary sarcoidosis. This study investigated the safety and efficacy of 10 mg/kg CMK389 administered intravenously (i.v.) every 4 weeks for a total of 4 doses, versus placebo

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a body mass index (BMI) at screening within the range of 18 - 46 kg/m2. BMI = Body weight (kg) / [Height (m)]2
* Biopsy proven pulmonary sarcoidosis diagnosed > 1 year prior to screening
* Scadding stage II, III or IV as determined by the most recent chest x-ray obtained within 12 months prior to screening or at screening (confirmed by the Investigator)
* HRCT extent of fibrosis <20% (confirmed by the central imaging reader) at screening
* Treatment with 5-15 mg/day prednisone (or prednisone oral equivalents) for ≥ 6 months prior to screening.
* Co-medication with methotrexate or azathioprine for ≥ 6 months prior to screening (Note: hydroxychloroquine is allowed as background therapy but not required)
* Able to perform reliable, reproducible pulmonary function test maneuvers per American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines

Exclusion Criteria:

* Diagnosis of significant pulmonary hypertension (WHO group 5) requiring pharmacological treatment
* Active cardiac sarcoidosis requiring treatment. Inactive cardiac sarcoidosis or stable cardiac sarcoidosis not requiring treatment are permissible.
* A known diagnosis of neurosarcoidosis
* Forced vital capacity (FVC) <50% of predicted at screening (central read)
* Modified British Medical Research Council (mMRC) dyspnea scale ≥ 3 at screening
* Concomitant treatment with leflunomide, cyclophosphamide, mycophenolate, infliximab, etanercept, adalimumab, golimumab, ustekinumab, roflumilast, pentoxifylline, and abatacept within 12 weeks of screening
* Prior treatment with rituximab, canakinumab, anakinra, and tocilizumab
* Current use of any inhaled substance, including but not limited to tobacco, marijuana products and use of electronic cigarette or vaping device, and excluding inhalers or nebulizers prescribed for pulmonary sarcoidosis
* Any conditions or significant medical problems which in the opinion of the investigator and in consultation with the sponsor, immunocompromises the patient and/or places the patient at unacceptable risk for immunomodulatory therapy
* Contraindication to FDG-PET scan investigations such as severe claustrophobia or uncontrolled diabetes
* History or current diagnosis of ECG abnormalities not due to Cardiac Sarcoidosis and indicating significant risk of safety for patients participating in the study
* A diagnosis of Lofgren's syndrome
* A history of pancreatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - Novartis Investigative Site, Birmingham, Alabama
  - Univ of Florida College of Medicine x, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - John Hopkins Asthma And Alrgy Cntr, Baltimore, Maryland
  - Icahn School Of Med At Mount Sinai ., New York, New York
  - East Carolina University ., Greenville, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
- Denmark (3):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Hellerup
  - Novartis Investigative Site, Odense C
- Germany (5):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Warsaw
- United Kingdom (2):
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 22 investigative sites in 6 countries.
Pre-assignment Details: After obtaining signed informed consent, a screening epoch of 28 days was used to assess subject eligibility.
Groups:
- CMK389 10 mg/kg i.v.: CMK389 10 mg/kg i.v. every 4 weeks for a total of 4 doses
- Placebo i.v.: Placebo i.v. every 4 weeks for a total of 4 doses
Period: Overall Study
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v. | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (8.69) | 50.7 (9.36) | 51.1 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 24 | 18 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 3 | 2 | 5
  Unknown | 0 | 1 | 1
  White | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Predicted FVC From Baseline to 16 Weeks of Treatment
Description: To assess the effect of CMK389 compared to placebo after 16 weeks of treatment on spirometry (Forced Vital Capacity). Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Percent predicted FVC is the percentage of the age, height and gender adjusted predicted value.
Time Frame: Baseline, Week 16
Population: The Pharmacodynamic (PD) analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data. Data collected after a change of the steroid dose not based on the clinical status evaluation (CSE) algorithm were excluded from the analysis set if assessed as having a potentially relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 26 | 27
Percent predicted | -0.48 (1.17) | 1.02 (1.13)
Statistical Analysis 1: Comparison: CMK389 10 mg/kg i.v. vs Placebo i.v; Test type: Other — A Bayesian model for repeated measurements including data collected at Weeks 4, 8, 12 and 16 was applied to compare FVC between CMK389 and placebo groups; p = 0.1804, Bayesian analysis; Posterior probability that treatment is better than placebo; Posterior estimate treatment difference = -1.49, 80% CI 2-sided [-3.56 to 0.60], Standard Deviation 1.62 — 80% credible intervals are reported on the treatment difference

2. Secondary Outcome: Number of Participants Who Had an Increase in Steroid Usage From Baseline to 16 Weeks of Treatment
Description: The Clinical Status Evaluation (CSE) served as a safety evaluation and served to establish the patient's clinical status (Clinical Status Determination [CSD]). CSE was performed prior to the titration of steroids, and the CSD guided selection of the next dose of steroids. Participants with CSD of "improved" or "stable" decreased steroid dose by 1 step on the dosing scale. Participants with CSD of "deteriorating" were ineligible to continue the study (if found during the run-in epoch or at study Day 1); or they increased steroid dose by 1 step (if found during the treatment epoch).
Time Frame: Baseline, Week 16
Population: The PD analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data. Data collected after a change of the steroid dose not based on the CSE algorithm were excluded from the analysis set if assessed as having a potentially relevant impact on PD data.
Measure: Count of Participants; unit: Participants
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 29 | 31
Participants | 5 | 4

3. Secondary Outcome: Number of Participants Who Deteriorate From Baseline to 16 Weeks of Treatment
Description: Composite index of pulmonary physiology (CIPP) and exercise capacity: a participant who deteriorated from baseline to each visit was defined as a patient with:
  relative reduction if FVC ≥ 10%, or relative reduction if FEV1 ≥ 10%, or relative reduction of DLCO ≥ 15%, or relative reduction of 6MWD ≥ 50 m.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 29 | 31
Participants | 9 | 10

4. Secondary Outcome: Percent Change in [18F]-FDG-PET/CT (SUVmax and SUVmean) From Baseline to 16 Weeks of Treatment
Description: [18F]-fluorodeoxyglucose positron emission tomography/computed tomography (FDG-PET/CT) maximum standardized uptake value and mean standardized uptake value (SUVmax and SUVmean) imaging was used to assess potential anti-inflammatory effects by CMK389 on the sarcoidosis process. All participants underwent whole-body head to mid-thigh [18F]FDG-PET/CT imaging state-of-the-art, 3D PET/CT scanners with a reconstructed resolution of ≤5 mm.
Time Frame: Baseline, Week 16
Population: The PD analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data. Data collected after a change of the steroid dose not based on the CSE algorithm were excluded from the analysis set if assessed as having a potentially relevant impact on PD data. This analysis included only participants with a baseline positron emission tomography (PET) signal in the corresponding region.
Measure: Least Squares Mean (Standard Error); unit: percent change from Baseline
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 29 | 31
percent change from Baseline
  Lung Parenchyma SUVmax: number analyzed (Participants) | 12 | 18
  Lung Parenchyma SUVmax | -29.23 (31.128) | 26.78 (24.461)
  Lymph Nodes SUVmax: number analyzed (Participants) | 11 | 9
  Lymph Nodes SUVmax | -23.40 (9.083) | -16.48 (9.759)
  Extrathoracic SUVmax: number analyzed (Participants) | 4 | 13
  Extrathoracic SUVmax | -12.89 (14.361) | -19.07 (6.908)
  Lung Parenchyma SUVmean: number analyzed (Participants) | 12 | 18
  Lung Parenchyma SUVmean | -34.06 (28.626) | 20.74 (22.443)
  Lymph Nodes SUVmean: number analyzed (Participants) | 11 | 9
  Lymph Nodes SUVmean | -30.83 (8.157) | -22.75 (9.101)
  Extrathoracic SUVmean: number analyzed (Participants) | 4 | 13
  Extrathoracic SUVmean | -11.23 (13.020) | -23.99 (6.440)

5. Secondary Outcome: The Observed Serum Concentration Following CMK389 Administration at End of Infusion
Description: Pharmacokinetic parameters were directly derived from the PK concentration data using non-compartmental analysis.
Time Frame: Post 1 hour: Day 1, Day 29, Day 57, Day 85
Population: The Pharmacokinetics (PK) analysis set included all patients with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received CMK389 and with no protocol deviations with relevant impact on PK data.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | CMK389 10 mg/kg i.v.
Number analyzed (Participants) | 31
ng/mL
  Day 1: number analyzed (Participants) | 30
  Day 1 | 453000 [236000 to 1230000]
  Day 29 | 533000 [58100 to 2460000]
  Day 57: number analyzed (Participants) | 29
  Day 57 | 571000 [77600 to 3070000]
  Day 85: number analyzed (Participants) | 28
  Day 85 | 541000 [78300 to 893000]

6. Secondary Outcome: Pre-dose Trough Concentration (Ctrough) of CMK389
Description: Pharmacokinetic parameters were directly derived from the PK concentration data using non-compartmental analysis. Ctrough is the observed plasma concentration that is just prior to the beginning of a dosing interval.
Time Frame: Pre-dose: Day 1, Day 29, Day 57, Day 85
Population: The PK analysis set included all patients with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received CMK389 and with no protocol deviations with relevant impact on PK data.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | CMK389 10 mg/kg i.v.
Number analyzed (Participants) | 31
ng/mL
  Day 1: number analyzed (Participants) | 15
  Day 1 | 0.00 [0.00 to 619000]
  Day 29 | 83500 [43300 to 176000]
  Day 57: number analyzed (Participants) | 30
  Day 57 | 105000 [41700 to 182000]
  Day 85: number analyzed (Participants) | 30
  Day 85 | 125000 [27900 to 444000]

7. Secondary Outcome: Change in FEV1 From Baseline to 16 Weeks of Treatment
Description: FEV1 (forced expiratory volume in one second) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The least-squares means for change from baseline in FEV1 to assess the effect of CMK389 compared to placebo after 16 weeks were obtained from a mixed effects model for repeated measures (MMRM). A positive change from baseline in pre-dose FEV1 is considered a favourable outcome.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters (L)
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 26 | 27
liters (L) | -0.03 (0.033) | 0.00 (0.032)
Statistical Analysis 1: Comparison: CMK389 10 mg/kg i.v. vs Placebo i.v; Test type: Superiority; p = 0.783, Mixed effects Model for Repeated Measure; Median Difference (Net) = -0.04, 80% CI 2-sided [-0.09 to 0.02], Standard Error of Mean 0.045 — Treatment difference (CMK389-placebo)

8. Secondary Outcome: Change in Diffusion Capacity of the Lung for Carbon Monoxide (DLCO) From Baseline to 16 Weeks of Treatment
Description: DLCO is a measurement to assess the lungs' ability to transfer gas from inspired air to the bloodstream. The least squares means for change from baseline in DLCO to assess the effect of CMK389 compared to placebo after 16 weeks were obtained from a mixed effects model for repeated measures (MMRM). A positive change from baseline in DLCO is considered a favourable outcome.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mL/min/mmHg
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 20 | 25
mL/min/mmHg | -0.58 (0.493) | -0.40 (0.448)
Statistical Analysis 1: Comparison: CMK389 10 mg/kg i.v. vs Placebo i.v; Test type: Superiority; p = 0.608, Mixed effects Model for Repeated Measure; Mean Difference (Net) = -0.18, 80% CI 2-sided [-1.05 to 0.68], Standard Error of Mean 0.664 — Treatment difference (CMK389-placebo)

9. Secondary Outcome: Change in 6-minute Walk Distance (6MWD) From Baseline to 16 Weeks of Treatment
Description: The 6MWD test is self-paced, with standardized instructions and encouragement being given as participants walk as far as possible over 6 minutes through a flat corridor. The final distance is recorded in meters. The least squares means for change from baseline in 6MWD to assess the effect of CMK389 compared to placebo after 16 weeks were obtained from a mixed effects model for repeated measures (MMRM). A positive change from baseline in 6MWD is considered a favourable outcome.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | CMK389 10 mg/kg i.v. | Placebo i.v.
Number analyzed (Participants) | 26 | 26
meters | 11.21 (9.470) | 10.50 (9.223)
Statistical Analysis 1: Comparison: CMK389 10 mg/kg i.v. vs Placebo i.v; Test type: Superiority; p = 0.479, Mixed effects Model for Repeated Measure; Median Difference (Net) = 0.71, 80% CI 2-sided [-16.35 to 17.76], Standard Error of Mean 13.126 — Treatment difference (CMK389-placebo)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 197 days..
Groups:
- Total: Total
Arm/Group | CMK389 10 mg/kg i.v | Placebo i.v | Total
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/62
Serious Adverse Events (participants affected / at risk) | 2/31 | 0/31 | 2/62
Other Adverse Events (participants affected / at risk) | 21/31 | 19/31 | 40/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMK389 10 mg/kg i.v (N=31) | Placebo i.v (N=31) | Total (N=62)
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CMK389 10 mg/kg i.v (N=31) | Placebo i.v (N=31) | Total (N=62)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 3 | 1 | 4
Chest pain (General disorders) | 3 | 1 | 4
Fatigue (General disorders) | 4 | 4 | 8
COVID-19 (Infections and infestations) | 3 | 4 | 7
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 6
Urinary tract infection (Infections and infestations) | 1 | 3 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 2
Blood creatinine increased (Investigations) | 2 | 0 | 2
Lipase increased (Investigations) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Dizziness (Nervous system disorders) | 3 | 1 | 4
Headache (Nervous system disorders) | 2 | 4 | 6
Haematuria (Renal and urinary disorders) | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Cutaneous sarcoidosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Hypertension (Vascular disorders) | 2 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT04064242/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT04064242/SAP_001.pdf